CLINICAL TRIAL: NCT04748523
Title: Effect of Mirtazapine Versus Placebo on Appetite, Nutritional Status and Quality of Life in Non-small Cell Lung cáncer Patients With Anorexia; Randomized Double-blind Clinical Trial.
Brief Title: Effect of Mirtazapine Versus Placebo in Patients With Non-small Cell Lung Cancer and Anorexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, M.D.,M.Sc., Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mirtazapine
Record Dates: First submitted 2020-11-19; First posted 2021-02-10 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Anorexia; Non-small Cell Lung Cancer
MeSH Terms: conditions — Anorexia; Carcinoma, Non-Small-Cell Lung | interventions — Mirtazapine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Mirtazapine and placebo containers of same appearance will be identified with a code, which will be uncovered at the end of the study. The codes assigned to Mirtazapine and placebo will be protected by the protocols coordination of the Functional Unit of Thoracic Oncology. The code will be assigned to patients in order of admission, according to a list pre-established by random numbers without knowing to which group the attending physician, the nutritionist, the psychiatrist or the patient belongs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): arm to receive 15 to 30 mg of Mirtazapine for a period of 8 weeks.
  Interventions: Drug: Mirtazapine
- Placebo group (Placebo Comparator): arm to receive 15 to 30 mg of placebo for a period of 8 weeks.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Mirtazapine — arm to receive 15 to 30 mg of Mirtazapine for a period of 8 weeks.
  Arms: Intervention group
Drug: Placebo Oral Tablet — arm to receive 15 to 30 mg of Placebo for a period of 8 weeks.
  Other Names: Placebo
  Arms: Placebo group

SUMMARY:
The realization of this project will generate an important advance in knowledge regarding one of the most important comorbidities in cancer patients: malnutrition.

Currently, comprehensive treatments of cancer patients recognize the importance of the assessment of nutritional status, and the impact it has on the prognosis, quality of life and toxicity generated by cancer treatment. Due to this, it is imperative to offer diagnostic tools that identify patients in a timely manner and, in addition to this, offer therapeutic strategies for the improvement of nutritional status, in an adjuvant manner to their oncological treatment.

It is widely recognized that the cachexia-anorexia syndrome (CACS) is present in 30 to 80% of cases in cancer patients and this proportion increases as the disease progresses, with weight loss being a powerful predictor of shorter survival. Unfortunately, current therapies available to treat anorexia and / or cancer-associated cachexia offer only partial results, mainly because the intervention is late and the development of an earlier and more effective intervention is still sought. Mirtazapine has recently gained attention not only because of its antidepressant effect, but also because of its potential benefit in patients with anorexia and weight loss, recently reported in a phase II study. Therefore, it is important to continue its evaluation through a randomized, double-blind clinical trial in which the effect of mirtazapine is compared and it is determined if it is superior compared to placebo to increase appetite in patients with NSCLC who present with anorexia.

This type of strategy is a relevant therapeutic option in those patients in whom nutritional counseling by itself is not sufficient to counteract the damage caused by anorexia and to cope with or prevent the development of cachexia.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in Mexico and the world. One of the comorbidities most commonly associated with this type of malignancy is malnutrition, which occurs in approximately 40-50% of newly diagnosed cases. In addition to its high incidence, malnutrition in patients with cancer is of great relevance due to the negative effect that this entails on the quality of life and the prognosis of patients, as well as the increase in toxicity associated with oncological treatment. Malnutrition is a pathological state in which the deficiency in the adequate contribution of energy contributes to its development, producing a systemic catabolic state; Its etiology is variable, however, in most patients malnutrition is associated with a lack of appetite, which is called anorexia.

Mirtazapine is a tetracyclic antidepressant which has been widely used for the treatment of depression. Several clinical studies have proven its efficacy in this indication, with more than 5000 patients endorsing its clinical effect compared to placebo, other tetracyclic antidepressants and trazodone. In addition to its effect on mood, it has been observed that mirtazapine, used in standard doses, induces weight gain, increasing appetite and food consumption compared to patients receiving placebo.

The increase in appetite with consequent weight gain and increased food intake may be due to the blocking of 5HT1b, 5-HT2, 5-HT3, H1 receptors, involved in the regulation of appetite. A pilot study of 2 doses of mirtazapine (15 or 30 mg per day) in ambulatory cancer patients with pain and other discomforts suggests that it provides a significant improvement in quality of life, particularly in weight and energy intake. Recently, another phase II study observed that 57% of oncology patients, ambulatory, non-depressed, increased their appetite and body weight when treated with mirtazapine for 4 weeks. Despite these encouraging data, the study included a small sample of patients, so it is not possible to generate robust conclusions from these data.

The objective of this protocol is to conduct a prospective, randomized, double-blind clinical trial to evaluate the effect of Mirtazapine on appetite, nutritional status and quality of life in patients with anorexia associated with lung cancer. The sample would include 86 patients, 43 patients with Mirtazapine and 43 sith placebo for 8 weeks, with an inducing dose of 15 mg to a máximum of 30 mg. The methodology for conducting this study consists of recruiting patients diagnosed with anorexia according to the anorexia-cachexia (ACS) scale, which has a cut-off point specifically validated for lung cáncer. Once the patient is selected, they are invited to participate in the study and an informed consent is requested. Subsequently a subjective global evaluation is performed, a 24-hour reminder of energy consumption, evaluation of anthropometric measures (weight, height,% weight loss, body mass index), evaluation of body composition (% fat, fat-free mass and phase angle), common gastrointestinal adverse effects of chemotherapy according to CTCAE, an evaluation of anxiety and depression (HADS) , as well as determination of quality of life through the questionnaire "The European organization for research and treatment of cancer quality of life questionnaire (QLQ) -C30 and (QLQ) LC-13", validated for Mexican population.

All determinations will be made at baseline, at 4 and at 8 weeks. All the variables are going to be evaluated inside each groups and between groups. It´s going to be considered significant p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients over 18 years of age who are receiving care in INCan with histopathological diagnosis of advanced stage non-small cell lung cancer (IIIB or IV).
* A score ≤ 32 on the cachexia anorexia scale or ≥ 5% weight loss in the last month.
* Good performance status (ECOG 0-2)
* That they are receiving chemotherapy as standard treatment or tyrosine kinase inhibitors or immunotherapy.
* Have a life expectancy> 8 weeks.
* Accept and sign informed consent letter.

Exclusion Criteria:

* Known allergy to mirtazapine
* Patients who are treated with antidepressants
* Patients who are under treatment with megestrol acetate
* Patients with moderate hepatic and / or renal dysfunction (bilirubin level ≥ 1.5 x above normal limits (UNL), AST and ALT ≥ 5 x UNL, or creatinine ≥5 x UNL).
* Those unable to take medication orally.
* Patients with mechanical obstruction of the gastrointestinal tract, ascites or generalized edema.
* Patients with a history of phenylketonuria (preparation contains phenylalanine).
* Patients with delirium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — adults
Enrollment: 86 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-10-29 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with Anorexia | From the baseline assessment to 4 and 8 weeks
  The primary endpoint will assess the percentage of patients who continue to present anorexia after 4 and 8 weeks of treatment with placebo or mirtazapine.
  Anorexia will be defined as the lack of desire to eat, lack of appetite, as measured using the validated version of the Anorexia / Cachexia Scale from the Functional Assessment of Anorexia Cachexia Therapy (FAACT). A score of less than or equal to 24 will be considered diagnostic for anorexia.
Energy Consumption | From the baseline assessment to 4 and 8 weeks
  Total kilocalories consumed on average per day by a subject

SECONDARY OUTCOMES:
Weight | From the baseline assessment to 8 weeks
  Sum of all the components of the organism and represents the total body mass.
Body Mass Index | From the baseline assessment to 8 weeks
  It is an index of the weight of a person in relation to his height BMI = Weight (Kg.) / [height (m) * height) (m)]
Subjetive Global Assessment | From the baseline assessment to 8 weeks
  Practical, quick and lower cost method used to make a nutritional evaluation, which consists of 3 parts: Anamnesis, physical examination and qualification.
  A: Patients with an adequate nutritional status B: Suspected malnutrition or moderate malnutrition C: Patients with severe malnutrition
Protein consumption | From the baseline assessment to 8 weeks
  Grams of protein consumed on average per day by a subject
Lipids consumption | From the baseline assessment to 8 weeks
  Grams of lipids consumed on average per day by a subject
Carbohydrates consumption | From the baseline assessment to 8 weeks
  Grams of carbohydrates consumed on average per day by a subject
Body fat | From the baseline assessment to 8 weeks
  Body fat
Fat free mass | From the baseline assessment to 8 weeks
  skeletal muscle, visceral protein, plasma proteins, extracellular water, skin and skeleton.
phase angle | From the baseline assessment to 8 weeks
  Angular transformation of the ratio of reactance to resistance
Quality of life - Global status | From the baseline assessment to 8 weeks
  Physical, physiological and social factors in the life of a patient. The Global status of Quality of Life evaluation will be evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer (EORTC) Quality of life questionnaires specific for cancer with the items 29 and 30 (QLQ-C30 version 3.0) and complemented with the quality of life questionnaire for lung cancer (QLQ-LC13).
  Scores range from 0-100, with higher scores representing better quality of life.
  The items included in each scale are calculated a raw count (average = s score) and the corresponding formula is applied to obtain the final count (Score).
Quality of life - physical functioning | From the baseline assessment to 8 weeks
  The physical functioning will be evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer (EORTC) Quality of life questionnaires specific for cancer using the physical functioning scale (from QLQ-C30 version 3.0).
  Scores range from 0-100, with higher scores representing better physical functioning.
  The items included in each scale are calculated a raw count (average = s score) and the corresponding formula is applied to obtain the final count (Score).
Quality of life -Role functioning | From the baseline assessment to 8 weeks
  The role functioning will be evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer (EORTC) Quality of life questionnaires specific for cancer using the role functioning scale (from QLQ-C30 version 3.0).
  Scores range from 0-100, with higher scores representing better role functioning.
  The items included in each scale are calculated a raw count (average = s score) and the corresponding formula is applied to obtain the final count (Score).
Quality of life - Emotional functioning | From the baseline assessment to 8 weeks
  The emotional functioning will be evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer (EORTC) Quality of life questionnaires specific for cancer using the emotional functioning scale (from QLQ-C30 version 3.0).
  Scores range from 0-100, with higher scores representing better emotional functioning.
  The items included in each scale are calculated a raw count (average = s score) and the corresponding formula is applied to obtain the final count (Score).
Quality of life - Cognitive functioning | From the baseline assessment to 8 weeks
  The cognitive functioning will be evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer (EORTC) Quality of life questionnaires specific for cancer using the cognitive functioning scale (from QLQ-C30 version 3.0).
  Scores range from 0-100, with higher scores representing better cognitive functioning.
  The items included in each scale are calculated a raw count (average = s score) and the corresponding formula is applied to obtain the final count (Score).
Quality of life - Social functioning | From the baseline assessment to 8 weeks
  The social functioning will be evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer (EORTC) Quality of life questionnaires specific for cancer using the social functioning scale (from QLQ-C30 version 3.0).
  Scores range from 0-100, with higher scores representing better social functioning.
  The items included in each scale are calculated a raw count (average = s score) and the corresponding formula is applied to obtain the final count (Score).
Quality of life - Fatigue | From the baseline assessment to 8 weeks
  Fatigue will be evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer (EORTC) Quality of life questionnaires specific for cancer using the fatigue symptom scale (from QLQ-C30 version 3.0).
  Scores range from 0-100, with higher scores representing worse fatigue. The items included in each scale are calculated a raw count (average = s score) and the corresponding formula is applied to obtain the final count (Score).
Quality of life - Nausea and vomiting | From the baseline assessment to 8 weeks
  Nausea and vomiting will be evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer (EORTC) Quality of life questionnaires specific for cancer using the nausea and vomiting symptom scale (from QLQ-C30 version 3.0).
  Scores range from 0-100, with higher scores representing worse nausea and vomiting.
  The items included in each scale are calculated a raw count (average = s score) and the corresponding formula is applied to obtain the final count (Score).
Quality of life - loss of appetite | From the baseline assessment to 8 weeks
  Loss of appetite will be evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer (EORTC) Quality of life questionnaires specific for cancer using the loss of appetite single item (from QLQ-C30 version 3.0).
  Scores range from 0-100, with higher scores representing worse loss of appetite.
  The items included in each scale are calculated a raw count (average = s score) and the corresponding formula is applied to obtain the final count (Score).
Anxiety | From the baseline assessment to 8 weeks
  Mental state characterized by great restlessness, intense excitement and extreme insecurity.
  Anxiety will be evaluated using the Mexican version of the Hospital Anxiety and Depression Scale (HADS) which was validated by Galindo Vázquez et al. (2015) is comprised of a scale which includes 14 items, which have four options as answers (ranging from 0-3). Scores range from 0-21. Highest scores denote higher anxiety.
Depression | From the baseline assessment to 8 weeks
  Illness or mental disorder that is characterized by a deep sadness, mood decay, low self-esteem, loss of interest in everything and decrease in psychic functions. Depression will be evaluated using the Mexican version of the Hospital Anxiety and Depression Scale (HADS) which was validated by Galindo Vázquez et al. (2015) is comprised of a scale which includes 14 items, which have four options as answers (ranging from 0-3). Scores range from 0-21. Highest scores denote higher depression.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G Arrieta Rodriguez, M.D., M.Sc., Principal Investigator — Instituto Nacional de Cancerología de México
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Watanabe H, Yamamoto N, Tamura T, Shimoyama T, Hotta K, Inoue A, Sawada M, Akiyama Y, Kusaba H, Nokihara H, Sekine I, Kunitoh H, Ohe Y, Kodama T, Saijo N. Study of paclitaxel and dose escalation of cisplatin in patients with advanced non-small cell lung cancer. Jpn J Clin Oncol. 2003 Dec;33(12):626-30. doi: 10.1093/jjco/hyg116. PMID 14769840
- [Background] Sarhill N, Mahmoud FA, Christie R, Tahir A. Assessment of nutritional status and fluid deficits in advanced cancer. Am J Hosp Palliat Care. 2003 Nov-Dec;20(6):465-73. doi: 10.1177/104990910302000610. PMID 14649565
- [Background] Arrieta O, Michel Ortega RM, Villanueva-Rodriguez G, Serna-Thome MG, Flores-Estrada D, Diaz-Romero C, Rodriguez CM, Martinez L, Sanchez-Lara K. Association of nutritional status and serum albumin levels with development of toxicity in patients with advanced non-small cell lung cancer treated with paclitaxel-cisplatin chemotherapy: a prospective study. BMC Cancer. 2010 Feb 21;10:50. doi: 10.1186/1471-2407-10-50. PMID 20170547
- [Background] Sanchez-Lara K, Turcott JG, Juarez E, Guevara P, Nunez-Valencia C, Onate-Ocana LF, Flores D, Arrieta O. Association of nutrition parameters including bioelectrical impedance and systemic inflammatory response with quality of life and prognosis in patients with advanced non-small-cell lung cancer: a prospective study. Nutr Cancer. 2012;64(4):526-34. doi: 10.1080/01635581.2012.668744. Epub 2012 Apr 10. PMID 22489794
- [Background] Wie GA, Cho YA, Kim SY, Kim SM, Bae JM, Joung H. Prevalence and risk factors of malnutrition among cancer patients according to tumor location and stage in the National Cancer Center in Korea. Nutrition. 2010 Mar;26(3):263-8. doi: 10.1016/j.nut.2009.04.013. Epub 2009 Aug 8. PMID 19665873
- [Background] Ross PJ, Ashley S, Norton A, Priest K, Waters JS, Eisen T, Smith IE, O'Brien ME. Do patients with weight loss have a worse outcome when undergoing chemotherapy for lung cancers? Br J Cancer. 2004 May 17;90(10):1905-11. doi: 10.1038/sj.bjc.6601781. PMID 15138470
- [Background] Slaviero KA, Read JA, Clarke SJ, Rivory LP. Baseline nutritional assessment in advanced cancer patients receiving palliative chemotherapy. Nutr Cancer. 2003;46(2):148-57. doi: 10.1207/S15327914NC4602_07. PMID 14690790
- [Background] Muscaritoli M, Anker SD, Argiles J, Aversa Z, Bauer JM, Biolo G, Boirie Y, Bosaeus I, Cederholm T, Costelli P, Fearon KC, Laviano A, Maggio M, Rossi Fanelli F, Schneider SM, Schols A, Sieber CC. Consensus definition of sarcopenia, cachexia and pre-cachexia: joint document elaborated by Special Interest Groups (SIG) "cachexia-anorexia in chronic wasting diseases" and "nutrition in geriatrics". Clin Nutr. 2010 Apr;29(2):154-9. doi: 10.1016/j.clnu.2009.12.004. Epub 2010 Jan 8. PMID 20060626
- [Background] Marin Caro MM, Laviano A, Pichard C. Impact of nutrition on quality of life during cancer. Curr Opin Clin Nutr Metab Care. 2007 Jul;10(4):480-7. doi: 10.1097/MCO.0b013e3281e2c983. PMID 17563467
- [Background] Kosacka M, Werynska B, Golecki M, Jankowska R, Passowicz-Muszynska E. [The incidence and pathogenesis of cancer anorexia-cachexia syndrome in lung cancer]. Pneumonol Alergol Pol. 2008;76(5):360-5. Polish. PMID 19003767
- [Background] Laviano A, Meguid MM, Inui A, Muscaritoli M, Rossi-Fanelli F. Therapy insight: Cancer anorexia-cachexia syndrome--when all you can eat is yourself. Nat Clin Pract Oncol. 2005 Mar;2(3):158-65. doi: 10.1038/ncponc0112. PMID 16264909
- [Background] Dewys WD, Begg C, Lavin PT, Band PR, Bennett JM, Bertino JR, Cohen MH, Douglass HO Jr, Engstrom PF, Ezdinli EZ, Horton J, Johnson GJ, Moertel CG, Oken MM, Perlia C, Rosenbaum C, Silverstein MN, Skeel RT, Sponzo RW, Tormey DC. Prognostic effect of weight loss prior to chemotherapy in cancer patients. Eastern Cooperative Oncology Group. Am J Med. 1980 Oct;69(4):491-7. doi: 10.1016/s0149-2918(05)80001-3. PMID 7424938
- [Background] Martin L, Senesse P, Gioulbasanis I, Antoun S, Bozzetti F, Deans C, Strasser F, Thoresen L, Jagoe RT, Chasen M, Lundholm K, Bosaeus I, Fearon KH, Baracos VE. Diagnostic criteria for the classification of cancer-associated weight loss. J Clin Oncol. 2015 Jan 1;33(1):90-9. doi: 10.1200/JCO.2014.56.1894. Epub 2014 Nov 24. PMID 25422490
- [Background] LeBlanc TW, Samsa GP, Wolf SP, Locke SC, Cella DF, Abernethy AP. Validation and real-world assessment of the Functional Assessment of Anorexia-Cachexia Therapy (FAACT) scale in patients with advanced non-small cell lung cancer and the cancer anorexia-cachexia syndrome (CACS). Support Care Cancer. 2015 Aug;23(8):2341-7. doi: 10.1007/s00520-015-2606-z. Epub 2015 Jan 14. PMID 25586527
- [Background] Gupta D, Lammersfeld CA, Vashi PG, King J, Dahlk SL, Grutsch JF, Lis CG. Bioelectrical impedance phase angle in clinical practice: implications for prognosis in stage IIIB and IV non-small cell lung cancer. BMC Cancer. 2009 Jan 28;9:37. doi: 10.1186/1471-2407-9-37. PMID 19175932
- [Result] Bossola M, Pacelli F, Doglietto GB. Novel treatments for cancer cachexia. Expert Opin Investig Drugs. 2007 Aug;16(8):1241-53. doi: 10.1517/13543784.16.8.1241. PMID 17685872
- [Result] Munzer A, Sack U, Mergl R, Schonherr J, Petersein C, Bartsch S, Kirkby KC, Bauer K, Himmerich H. Impact of antidepressants on cytokine production of depressed patients in vitro. Toxins (Basel). 2013 Nov 19;5(11):2227-40. doi: 10.3390/toxins5112227. PMID 24257035
- [Result] Langer CJ, Hoffman JP, Ottery FD. Clinical significance of weight loss in cancer patients: rationale for the use of anabolic agents in the treatment of cancer-related cachexia. Nutrition. 2001 Jan;17(1 Suppl):S1-20. doi: 10.1016/s0899-9007(01)80001-0. No abstract available. PMID 11428126
- [Result] Capra S, Ferguson M, Ried K. Cancer: impact of nutrition intervention outcome--nutrition issues for patients. Nutrition. 2001 Sep;17(9):769-72. doi: 10.1016/s0899-9007(01)00632-3. PMID 11527676
- [Result] Anttila SA, Leinonen EV. A review of the pharmacological and clinical profile of mirtazapine. CNS Drug Rev. 2001 Fall;7(3):249-64. doi: 10.1111/j.1527-3458.2001.tb00198.x. PMID 11607047
- [Result] Hilas O, Avena-Woods C. Potential role of mirtazapine in underweight older adults. Consult Pharm. 2014 Feb;29(2):124-30. doi: 10.4140/TCP.n.2014.124. PMID 24513422
- [Result] Kumar N, Barai S, Gambhir S, Rastogi N. Effect of Mirtazapine on Gastric Emptying in Patients with Cancer-associated Anorexia. Indian J Palliat Care. 2017 Jul-Sep;23(3):335-337. doi: 10.4103/IJPC.IJPC_17_17. PMID 28827942
- [Result] Lopez-Llera M. Eclampsia and fetal sex. Int J Gynaecol Obstet. 1990 Nov;33(3):211-3. doi: 10.1016/0020-7292(90)90003-4. PMID 1977637
- [Derived] Arrieta O, Cardenas-Fernandez D, Rodriguez-Mayoral O, Gutierrez-Torres S, Castanares D, Flores-Estrada D, Reyes E, Lopez D, Barragan P, Soberanis Pina P, Cardona AF, Turcott JG. Mirtazapine as Appetite Stimulant in Patients With Non-Small Cell Lung Cancer and Anorexia: A Randomized Clinical Trial. JAMA Oncol. 2024 Mar 1;10(3):305-314. doi: 10.1001/jamaoncol.2023.5232. PMID 38206631